CLINICAL TRIAL: NCT01052467
Title: Topical Treatment of Scalp Psoriasis With the Fixed Combination of Calcipotriol and Betamethason (Xamiol® Gel)
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: Treatment with Xamiol® Gel
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2010-09

CONDITIONS: Scalp Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Xamiol® Gel — Once daily application for about 4 weeks

SUMMARY:
This non-interventional, prospective, non-controlled study of Xamiol® Gel, a fixed combination of calcipotriol and betamethason dipropionate, shall investigate in daily routine the efficacy, tolerability and changes in quality-of-life parameters in patients with scalp psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Patients with scalp psoriasis if a treatment with Xamiol® gel is planned anyway

Exclusion Criteria:

* Contraindications of Xamiol® Gel listed in the German package insert
* Pretreatment with Xamiol® within the last 4 weeks
* Systemic treatment of psoriasis
* UV light therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visiting their attending dermatologist in the primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 724 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Physician's Global Assessment of scalp psoriasis | After approximately 4 weeks

SECONDARY OUTCOMES:
Patient's Quality of Life | After approximately 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Mrowietz, MD, Principal Investigator — University Clinic Schleswig-Holstein
Locations (1):
- University Clinical Schleswig-Holstein, Campus Kiel, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No